CLINICAL TRIAL: NCT03089320
Title: Financial Incentives, Randomization With Stepped Treatment Trial
Acronym: FIRST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: VA Connecticut Healthcare System (U.S. Federal Agency); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000020383; U01AA020795 (NIH)
Record Dates: First submitted 2017-03-17; First posted 2017-03-24 (Actual); Results first posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-03

CONDITIONS: Unhealthy Alcohol Use
Keywords: HIV, Heavy drinking, Alcohol Abuse, AIDS
MeSH Terms: conditions — Alcoholism; Acquired Immunodeficiency Syndrome | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment As Usual (TAU) (No Intervention): We have elected to compare the CM plus stepped care condition to TAU to test its efficacy against a "real world" control and because CM plus stepped care is a comprehensive stand alone intervention that would substitute for TAU. While annual AUDIT-C screening is mandatory at the 7 sites, providing interventions for patients with unhealthy alcohol use is a matter of physician judgment and individual clinical practice with wide practice variation. HIV clinicians will not receive knowledge of the results of follow-up research assessments. We will conduct a Treatment Services Review at each follow-up to assess for receipt of addiction treatment services received since the last assessment and assess for contamination.
- Contingency Management plus Stepped Care (Step 2) (Experimental): Step 1: Contingency management; Step 2: Addiction physician management and motivational enhancement therapy
  Consistent with tenets of stepped care designs we provide a priori intervals and criteria (drinking targets) that dictate increasing the intensity of treatment (stepping up) based on research and standards in the field. All CM plus stepped care subjects will undergo PEth testing at 3 months to determine the efficacy of Step 1. Patients with a PEth > 8 ng/ml will continue on to Step 2.
  Interventions: Behavioral: Contingency Management Counseling; Behavioral: Addiction Physician Management; Behavioral: Motivational Enhancement Therapy

INTERVENTIONS:
Behavioral: Contingency Management Counseling — Contingency management (CM) is an efficacious treatment for individuals with substance use disorders. In line with operant conditioning, CM typically provides reinforcers (rewards) contingent upon attaining specified goals such as decreased substance use and/or abstinence.
  Arms: Contingency Management plus Stepped Care (Step 2)
Behavioral: Addiction Physician Management — Patients in the CM plus stepped care arm who have PEth > 8 ng/ml at 3 months will progress to Step 2 and receive onsite treatment from an Addiction Psychiatrist (APM) in the HIV clinic. APM will provide care that is typically provided by physicians in specialty referral programs.
  Arms: Contingency Management plus Stepped Care (Step 2)
Behavioral: Motivational Enhancement Therapy — Patients in the CM plus stepped care arm who have PEth > 8 ng/ml at 3 months will progress to Step 2 and receive onsite Motivational Enhancement Therapy (MET) from the Social Worker in the HIV clinic.
  MET is grounded in research on processes of natural recovery during which patients move through stages of change - precontemplation, contemplation, determination, action, and maintenance. The Social Worker's role is to assist the patient in moving through the stages of change. MET uses motivational interviewing and reflective listening to help patients identify internal sources of motivation to support reductions in alcohol.
  Arms: Contingency Management plus Stepped Care (Step 2)

SUMMARY:
The investigators plan to determine the effectiveness of contingency management (CM) plus stepped care for unhealthy alcohol use in HIV-positive patients.

DETAILED DESCRIPTION:
HIV-positive patients with unhealthy alcohol use are not often motivated to decrease their alcohol consumption and rarely receive treatment for their drinking. To address these challenges, we plan to provide treatment in HIV clinics, highlight to patients the impact alcohol can have on their medical conditions, and use Contingency Management (CM) with a stepped care design to adjust treatment to patient response. CM is an evidence based therapy that promotes abstinence from substance use, including alcohol. Since CM has not been studied for unhealthy alcohol use in HIV-infected patients we will include a stepped care strategy that provides Addiction Psychiatrist Management (APM) (with alcohol pharmacotherapies as indicated) and Motivational Enhancement Therapy (MET) for patients who do not achieve abstinence with CM. Phosphatidylethanol (PEth), is a validated biomarker that can confirm alcohol abstinence over three weeks. To capture the range of adverse effects of alcohol on health, we will include patients with at-risk drinking, alcohol use disorder, and medical conditions that can be adversely impacted by alcohol including those with a detectable HIV viral load, tobacco use disorder, liver fibrosis, untreated hepatitis C, depression and those taking psychoactive medications that interact with alcohol. The goal of the Financial Incentives, Randomization with Stepped Treatment (FIRST) Trial is to compare onsite CM plus stepped care versus treatment as usual (TAU) in a randomized clinical trial of HIV-positive patients with unhealthy alcohol use at seven HIV clinics. CM patients will receive onsite CM counseling sessions with financial rewards contingent on abstinence demonstrated by breathalyzer and PEth. Rewards can also be awarded for addressing medical conditions impacted by alcohol and achieving alcohol treatment goals. After three months, patients will be stepped up to APM and MET if PEth results indicate they have not attained abstinence. This randomized clinical trial will test the hypothesis that CM plus stepped care leads to greater abstinence, decreased alcohol consumption and improved HIV biomarkers as measured by the VACS Index.

In addition to the randomized control trial, the FIRST Trial Implementation sub-study will be launched in the final year of the study. The goals of this sub-study are to explore barriers and facilitators to implementation of contingency management to address unhealthy alcohol in HIV treatment settings as it relates to: a) adoption, b) feasibility, c) acceptability, and d) tools and training needs to promote high fidelity implementation. In the context of the FIRST trial, we seek to recruit patient participants and the staff (i.e., research coordinators and Social Workers) involved with delivering CM across participating sites. Patient participants will be enrolled from the three highest-enrolling sites to complete an in-depth telephone interview. Staff participants from all sites involved in implementing study protocols will be invited to participate in a brief online survey and a focus group. Qualitative data will be analyzed by a multidisciplinary team using content analysis to identify themes and ideas regarding barrier and facilitators to CM implementation.

ELIGIBILITY:
Inclusion Criteria:

* Be HIV-infected.
* Recent significant alcohol consumption as determined by a PEth greater than 20 ng/ml.
* Able to provide informed consent.
* Meet any of the following criteria for unhealthy alcohol use:
* At-risk Drinking - greater than 14 drinks per week or greater than 4 drinks per occasion in men and greater than 7 drinks per week or greater than 3 drinks per occasion in women and those over 65.161
* Medical condition impacted by alcohol as evidenced by one of the following: 1) detectable HIV viral load (>200 copies/ml),) tobacco use disorder and smoking more than 5 cigarettes per day, 3) detectable HCV virus, 4) liver fibrosis with a FIB-4 >1.45) Patient Health Questionnaire (PHQ-9, validated measure for depression) score greater than 9, or 6) current (at least 30 day supply in the past 60 days) prescription for a psychoactive medication that interacts with alcohol-including benzodiazepines, opioids, antipsychotics, antidepressants, sleeping medications and muscle relaxants.
* Alcohol Use Disorder - Meet DSM-5 criteria for alcohol use disorder, not in remission

Exclusion Criteria:

No subject may:

* Be acutely suicidal, or with a psychiatric condition that affects his/her ability to provide informed consent or participate in counseling interventions (e.g. psychotic, dementia, delusional).
* Be currently enrolled in formal treatment for alcohol (excluding mutual-help, e.g. Alcoholics Anonymous)
* Have medical conditions that would preclude completing or be of harm during the course of the study.
* Be a pregnant or nursing woman or women who do not agree to use a reliable form of birth control.
* Have a current diagnosis of or be in remission for a gambling disorder given the gaming nature of CM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Fiellin, MD, Principal Investigator — Yale University; E. Jennifer Edelman, MD, Study Director — Yale University
Locations (7):
- United States (7):
  - Greater Los Angeles VA Healthcare Center Infectious Disease Section, Los Angeles, California
  - Washington DC Veterans Affairs, Washington D.C., District of Columbia
  - VA Medical Center, Atlanta, Georgia
  - Louisiana Health Sciences Center, New Orleans, Louisiana
  - VA NY Harbor Healthcare System, New York, New York
  - James J. Peters VA Medical Center, The Bronx, New York
  - VAMC Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edelman EJ, Dziura J, Deng Y, DePhilippis D, Ferguson T, Brown S, Marconi VC, Goetz MB, Rodriguez-Barradas MC, Simberkoff MS, Molina PE, Weintrob AC, Maisto SA, Paris M, Justice AC, Bryant KJ, Fiellin DA. Integrated Stepped Alcohol Treatment With Contingency Management for Unhealthy Alcohol Use Among People With HIV: A Randomized Controlled Trial. J Acquir Immune Defic Syndr. 2025 Jan 1;98(1):72-81. doi: 10.1097/QAI.0000000000003534. PMID 39321757
- [Derived] Edelman EJ, Dziura J, Deng Y, DePhilippis D, Fucito LM, Ferguson T, Bedimo R, Brown S, Marconi VC, Goetz MB, Rodriguez-Barradas MC, Simberkoff MS, Molina PE, Weintrob AC, Maisto SA, Paris M, Justice AC, Bryant KJ, Fiellin DA. Contingency management with stepped care for unhealthy alcohol use among individuals with HIV: Protocol for a randomized controlled trial. Contemp Clin Trials. 2023 Aug;131:107242. doi: 10.1016/j.cct.2023.107242. Epub 2023 May 23. PMID 37230168

RESULTS

PARTICIPANT FLOW:
Groups:
- Contingency Management Plus Stepped Care (Step 2): Step 1: Contingency management (CM); Step 2: Addiction physician management and motivational enhancement therapy We provide a priori intervals and criteria (drinking targets) that dictate increasing the intensity of treatment (stepping up) based on research and standards in the field. All CM plus stepped care subjects will undergo PEth testing at 3 months to determine the efficacy of Step 1. Patients with a PEth > 8 ng/ml will continue on to Step 2. Contingency Management Counseling: CM is an efficacious treatment for individuals with substance use disorders. In line with operant conditioning, CM provides reinforcers (rewards) contingent upon attaining specified goals such as decreased substance use and/or abstinence. Addiction Physician Management: Patients in the CM plus stepped care arm who have PEth > 8 ng/ml at 3 months will progress to Step 2 and receive onsite treatment from an Addiction Psychiatrist (APM) in the HIV clinic. APM will provide care that is typically provided by physicians in specialty referral programs. Motivational Enhancement Therapy: Patients in the CM plus stepped care arm who have PEth > 8 ng/ml at 3 months will progress to Step 2 and receive onsite MotivationalEnhancement Therapy (MET) from the Social Worker (SW) in the HIV clinic. The SW's role is to assist the patient in moving through the stages of change using motivational interviewing and reflective listening to help patients identify internal motivation to reduce alcohol use.
Period: Overall Study
Arm/Group | Treatment As Usual (TAU) | Contingency Management Plus Stepped Care (Step 2)
Started | 60 | 60
Completed | 57 | 51
Not Completed | 3 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment As Usual (TAU) | Contingency Management Plus Stepped Care (Step 2) | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.00 (8.29) | 58.65 (10.72) | 58.82 (9.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 59 | 56 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 13
  Not Hispanic or Latino | 50 | 50 | 100
  Unknown or Not Reported | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 53 | 47 | 100
  White | 6 | 9 | 15
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Abstinence From Alcohol
Description: Recorded via web based time-line followback
Time Frame: 6 months
Population: All participants randomized to CMSC orTAU.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Contingency Management Plus Stepped Care (Step 2) | Treatment As Usual (TAU)
Number analyzed (Participants) | 60 | 60
percentage of participants | 9.44 [0.1 to 32.89] | 0.32 [0 to 3.91]
Statistical Analysis 1: Comparison: Contingency Management Plus Stepped Care (Step 2) vs Treatment As Usual (TAU); Bayesian analysis was performed, therefore p value is not reported. Bayes factor has been reported instead; Test type: Superiority; posterior mean proportion of abstinence = 9.12, 95% CI 2-sided [0.08 to 31.68] — The lower and upper limits are credible intervals

2. Secondary Outcome: Proportion of Participants of Participants With Phosphatidylethanol (PeTH) Documented Abstinence by the Alcohol Biomarker, Phosphatidylethanol (PEth)
Description: Phosphatidylethanol (PEth) accumulates in human red blood cells when the body is exposed to ethanol. Alcohol biomarkers are physiological indicators of alcohol exposure or ingestion and may reflect the presence of chronic and/or high level of use of alcohol. This will be evaluated as a binary variable to determine the proportion with abstinence (defined as % with PEth value <8ng/mL).
Time Frame: 6 month
Population: All participants randomized to CMSC orTAU.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Contingency Management Plus Stepped Care (Step 2) | Treatment As Usual (TAU)
Number analyzed (Participants) | 60 | 60
percentage of participants | 5.86 [0.3 to 18.91] | 0.36 [0.00 to 3.59]
Statistical Analysis 1: Comparison: Contingency Management Plus Stepped Care (Step 2) vs Treatment As Usual (TAU); Bayesian analysis was performed, therefore p value is not reported. Bayes factor has been reported instead; Test type: Superiority; posterior mean proportion of abstinence = 5.5, 95% CI 2-sided [0.17 to 18.23] — The lower and upper limits are credible intervals

3. Secondary Outcome: Change in Biological Markers as Measured by the VACS Index
Description: The Veterans Aging Cohort Study Index (VACS Index) creates a score by summing pre-assigned points for age, routinely monitored indicators of HIV disease (CD4 count and HIV-1 RNA), and general indicators of organ system injury including hemoglobin, platelets, aspartate and alanine transaminase (AST and ALT), creatinine, and viral hepatitis C infection (HCV). This score is weighted to indicate increasing risk of all-cause mortality with increasing score. The score can be used to estimate risk of all-cause mortality using a conversion factor. The VACS Index will be evaluated based on most recent values at the time of data extraction. VACS Index score will be treated as a continuous variable. Possible scores range from 0 to 164. A higher score indicates greater burden of disease.
Time Frame: 6 months
Population: All participants randomized to CMSC or TAU
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Contingency Management Plus Stepped Care (Step 2) | Treatment As Usual (TAU)
Number analyzed (Participants) | 60 | 60
score on a scale | 30.25 [23.60 to 36.90] | 35.57 [27.46 to 41.68]
Statistical Analysis 1: Comparison: Contingency Management Plus Stepped Care (Step 2) vs Treatment As Usual (TAU); mixed effects model; Test type: Superiority; p = .05, Mixed Models Analysis; Mean Difference (Final Values) = -4.32, 95% CI 2-sided [-9.97 to 1.34], Standard Error of Mean 2.84

4. Other Pre Specified Outcome: Undetectable HIV Viral Load
Description: Viral load will be analyzed as a continuous measure (log10 copies/ml).
Time Frame: 6 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Smoking Cessation by Exhaled Carbon Monoxide
Description: It is measured by CO monitor
Time Frame: 6 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Liver Fibrosis Based on Fibrosis-4 (FIB-4) Score
Description: The Fibrosis-4 score helps to estimate the amount of scarring in the liver. Using a lower cutoff value of 1.45, a FIB-4 score <1.45 had a negative predictive value of 90% for advanced fibrosis (Ishak fibrosis score 4-6 which includes early bridging fibrosis to cirrhosis). In contrast, a FIB-4 >3.25 would have a 97% specificity and a positive predictive value of 65% for advanced fibrosis. In the patient cohort in which this formula was first validated, at least 70% patients had values <1.45 or >3.25.
Time Frame: 6 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Undetectable Hepatitis C Viral Load
Description: An HCV antibody test is used to screen for past exposure and current infection. It detects the presence of antibodies to the virus, indicating exposure to HCV.
Time Frame: 6 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Depressive Symptoms Via PHQ-9
Description: Patient Health Questionnaire (PHQ-9) ranges from 0 to 27. A higher score indicates worse depression. 5-9 are minimal symptoms, 10-14 is considered minor depression, 15-19 is major depression that is moderately severe, and >20 is severe, major depression.
Time Frame: 6 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Recent Receipt of a Psychoactive Medication That May Interact With Alcohol
Description: number of patients with use of psychoactive medications that interact with alcohol
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Treatment As Usual (TAU) | Contingency Management Plus Stepped Care (Step 2)
All-Cause Mortality (participants affected / at risk) | 0/60 | 2/60
Serious Adverse Events (participants affected / at risk) | 2/60 | 7/60
Other Adverse Events (participants affected / at risk) | 4/60 | 3/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment As Usual (TAU) (N=60) | Contingency Management Plus Stepped Care (Step 2) (N=60)
Death (General disorders) | 0 | 2 — Death, unrelated to study
Other SAEs (General disorders) | 1 | 5 — Other SAEs, organ system not reported
Respiratory SAE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment As Usual (TAU) (N=60) | Contingency Management Plus Stepped Care (Step 2) (N=60)
Other AE (General disorders) | 2 | 2 — Other AE, organ system not recorded
Psychiatric AE (Psychiatric disorders) | 2 | 0
Respiratory AE (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Respiratory adverse event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT03089320/Prot_SAP_001.pdf
  • Informed Consent Form (2021-02-27): https://cdn.clinicaltrials.gov/large-docs/20/NCT03089320/ICF_000.pdf